CLINICAL TRIAL: NCT02363049
Title: Randomized Phase III Study Assessing the Interest of Primary Tumor Resection in Patients With Asymptomatic Colon Cancer and Unresectable Synchronous Liver Metastases.
Brief Title: Colectomy in Patients With Asymptomatic and Unresectable Stage IV Colon Cancer
Acronym: CLIMAT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: UNICANCER (Other); Federation Francophone de Cancerologie Digestive (Other); GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-A00685-40
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Malignant Neoplasm of Large Intestine; Colon Cancer Liver Metastasis
Keywords: Colectomy; primary tumor resection; Asymptomatic primary colon cancer; Unresectable synchronous liver metastasis; TNM Staging Primary Tumor (T); Unresectable
MeSH Terms: conditions — Colonic Neoplasms | interventions — Colectomy; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- colectomy (Experimental): surgery followed by chemotherapy +/- targeted therapy regime according to each centre
  Interventions: Procedure: Colectomy; Drug: Chemotherapy
- no colectomy (Active Comparator): Chemotherapy +/- targeted therapy alone, regime according to each centre.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Procedure: Colectomy
  Arms: colectomy
Drug: Chemotherapy

SUMMARY:
The present study is a multicentric randomized phase III trial designed to assess whether overall survival and quality of life are improved in patients with asymptomatic colon cancer and unresectable SLM treated with resection of the PT followed by chemotherapy versus chemotherapy alone.

DETAILED DESCRIPTION:
At the time of diagnosis, 20-25% of patients with colorectal cancer (CRC) present synchronous liver metastases (SLM) and in the majority of patients (80-90%) liver metastases are unsuitable for curative surgical treatment. Whether either primary tumour (PT) resection followed by chemotherapy or immediate chemotherapy without PT resection is the best therapeutic option in patients with asymptomatic colon cancer and unresectable SLM is still controversial. No randomised trial has been conducted to answer this question.

Historically, surgeons have advocated resection of the PT to avoid potential complications of the intact PT (bleeding, obstruction, perforation). However, during the past decade, several highly active systemic agents have become available for treatment of patients with metastatic CRC. These agents have increased the median survival duration of patients with unresectable metastatic disease from 9 to 12 months with 5FU alone, to 30-35 months with the addition of modern cytotoxic and targeted agents. Modern agents have also demonstrated increased activity on the PT as well, and have been associated with low rates of PT-related complications during treatment in initially asymptomatic patients.

The impact of the strategy on survival has never been assessed properly. All published studies are of non-randomized design, single center, and retrospective in most of them. Moreover, few data on the use of systemic therapy are presented in these studies, which makes it difficult to assess the relative contribution of resection on outcome. In addition, patients with extensive disease or poor performance status were more likely to be offered chemotherapy rather than surgery thus introducing a bias at the ousted. Despite these limitations, PT resection at initial management of these metastatic CRC patients with unresectable SLM was related to prolonged survival on multivariate analysis in the majority of these series. The improvement in survival following PT resection may be attributed to the potential role of the PT to provide an angiogenic prosperous environment for metastatic tumour growth in the liver parenchyma adjacent to the SLM.

The present study is a multicenter randomized phase III trial designed to assess whether overall survival and quality of life are improved in patients with asymptomatic unresectable metastatic colon cancer treated with surgery followed by chemotherapy versus chemotherapy alone.

Patients (ECOG 0-1 performance status) with asymptomatic colon cancer (>15cm from the anal margin) and unresectable liver only metastatic disease on initial abdominal CT/MRI scan will be randomized to either colectomy followed by chemotherapy, or chemotherapy without resection of the PT. Systemic chemotherapy with or without targeted therapy will be let to the investigators' discretion according to standard local practices. The primary endpoint of the study is overall survival for >2 years. The secondary endpoints are: quality of life (EORTC QLQ-C30, QLQ-CR29), treatment safety (postoperative morbidity, complications related to the unresected PT, chemotherapy toxicity), progression-free survival and time to metastatic progression, radiological response to chemotherapy (RECIST v1.1 criteria), and the curative (R0) resection rate of metastases.

A 15% amelioration of overall survival at 2 years is expected in colectomy group (HR=0.65, with a rise from 40% to 55%). Using a two sided α level of 5%, 180 events are required to detect this difference with a power of 80% (β=0.20).

Taking into account the expected accrual of 15 patients per month during 19 months, a minimum follow-up of 28 months and a 5% rate of lost to follow-up, 278 patients will be included. The final analysis of all endpoints will be conducted 28 months after the last inclusion. The total duration of the study will be approximately 4 years.

A translational study will be conducted to evaluate the serum altered DNA patented test (AP-HP, 31 January 2008 under n°08/00543) we developed for colon cancer diagnosis, as a prognostic marker and a treatment response tool.

A radiological study will be conducted to identify the angiogenesis changes within or around liver metastases after resection of the PT. In addition to the morphological sequences allowing the use of RECIST1.1, DCE and DWI sequences will be performed in order to calculate the ADC value of the lesion as well as the Ktrans, Kep, PS that describe cellularity and perfusion of the lesions.

An optional ultrasound examination using SWE to study the stiffness of the liver metastases will be proposed at the end of the MRI examination.

ELIGIBILITY:
Inclusion criteria :

* Pathologically confirmed colon adenocarcinoma (≥ 15 cm from the anal verge)
* Uncomplicated PT (obstruction, bleeding, abcess, perforation)
* No known unresectable PT on CT/MRI scan.
* Unresectable synchronous liver metastases
* No extra-hepatic metastatic disease
* Age ≥ 18 years et ≤ 75 years
* ECOG performance status 0-1
* Life expectancy without cancer >2 years
* No prior chemotherapy in the past 5 years
* No prior abdominal or pelvic irradiation
* No history of colorectal cancer in the past 5years
* Patients with childbearing potential should use effective contraception during the study and the following 6 months
* White blood cell count ≥ 3 x 109/L with neutrophils ≥ 1.5 x 109/L, platelet count ≥ 100 x109/L, hemoglobin ≥ 9 g/dL (5,6 mmol/l)
* Total bilirubin <1.5 x ULN (upper limit of normal), ASAT and ALAT<2.5 x ULN, Alkaline phosphatase<1.5 x ULN, Serum creatinine < 1.5 x ULN
* Signed written informed consent obtained prior to any study specific screening procedures

Exclusion criteria :

* Resectable or potentially resectable liver metastases
* Complicated (obstruction, bleeding, abcess, perforation) or non resectable PT
* Rectal cancer located within 15 cm from the anal verge by endoscopy or under the peritoneal reflection at surgery or having received radiation therapy prior to surgery
* Age > 75 years
* ECOG performance status > 2
* Denutrition (albumin < 30 g/l)
* Synchronous colorectal cancer
* Extrahepatic metastatic disease
* Known hypersensitivity reaction or specific contraindications to any of the components of study treatments
* History of anti-EGFR or anti-VEGF treatment within the past 5 years
* History or current evidence on physical examination of central nervous system disease or
* peripheral neuropathy ≥ grade 1 Common Toxicity Criteria for Adverse Events (CTCAE) v.3.0
* Presence of inflammatory bowel disease
* HNPCC syndrome or polyposis
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to study treatment start. Incompletely healed wounds or anticipation of the need for major surgical procedure during the course of the study
* Clinically relevant coronary artery disease or history of myocardial infarction in the last 12 months, or high risk of uncontrolled arrhythmia
* Pregnancy (absence to be confirmed by ß-hCG test) or breast-feeding period
* Previous malignancy in the last 5 years
* Medical, geographical, sociological, psychological or legal conditions that would not permit the patient to complete the study or sign informed consent
* Any significant disease which, in the investigator's opinion, would exclude the patient from the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Estimated)
Dates: Start 2014-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
overall survival | 2 years

SECONDARY OUTCOMES:
quality of life | 2 years
  Questionnaire QLQ-C30 et QLQ-CR29 in both treatment arms Time frame : one month after surgery in arm A, one month after the beginning of chemotherapy in arm B and then each 3 months in both treatment arms up to 2 years
Post-operative complications | 30 days
  Post-operative complications (surgical or medical) will be graded according to the Clavien-Dindo system
Progression free survival (PFS) | 2 years
  PFS is defined as the time interval between the date of randomization and the first date of progression of the metastatic disease or death in both treatment arms.
  Time frame: each 3 months up to 2 years.
Time to metastatic progression (TTP) | 2 years
  TTP is defined as the time interval between the date of randomization and the first date of progression of the metastatic disease or death in both treatment arms in both treatment arms Time frame: each 3 months up to 2 years.
Rate of secondary curative resection (R0) | 1 year
  The rate of secondary curative resection will be assessed in both treatment arms and will concern resection of both the PT and the metastatic disease Time frame: each 3 months up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Karoui, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe hospitalier Pitié Salpetriere, Paris, France